CLINICAL TRIAL: NCT00951106
Title: Therapeutic Efficacy Study of Pyrimethamine / Sulfdoxine (Fansidar®) for the Treatment of Uncomplicated Falciparum Malaria in the Peruvian Amazon
Brief Title: Therapeutic Efficacy Study of Pyrimethamine/Sulfdoxine (Fansidar®) for the Treatment of Uncomplicated Falciparum Malaria in the Peruvian Amazon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: COL Alan Magill, WRAIR
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WRAIR #719
Record Dates: First submitted 2009-07-30; First posted 2009-08-04 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Malaria, Vivax; Malaria, Falciparum
Keywords: Peru; Sulfadoxine-pyrimethamine; Drug resistance
MeSH Terms: conditions — Malaria, Vivax; Malaria, Falciparum | interventions — Pyrimethamine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyrimethamine/sulfdoxine (Fansidar) (Experimental): Pyrimethamine/sulfdoxine (Fansidar)
  Interventions: Drug: Pyrimethamine/sulfdoxine (Fansidar)

INTERVENTIONS:
Drug: Pyrimethamine/sulfdoxine (Fansidar)

SUMMARY:
The purpose of this study is to determine the efficacy of pyrimethamine/sulfdoxine (Fansidar®) for the treatment of uncomplicated falciparum malaria in the Peruvian Amazon. Reports in the mid 1990s indicated that Fansidar was failing to cure patients with confirmed falciparum malaria. The study design was based on accepted WHO parasitological and clinical outcomes to determine the overall efficacy of Fansider and inform the Peruvian National Malaria Control authorities as to the continued wisdom of recommending Fansidar as first line treatment for uncomplicated falciparum malaria in the Peruvian Amazon.

ELIGIBILITY:
Inclusion Criteria:

* Pf monoinfection with asexual forms
* Parasite density of greater than 500 per mcl and less than 200 parasites per oil immersion field (MINSA quantification of "4 plus")
* Age > 6 months
* Temperature greater than 38C (101F)
* Available and willing to return for follow-up

Exclusion Criteria:

* Presence of any of the following "danger" signs or symptoms suggestive of severe malaria
* Not able to drink or breastfeed
* Repeated vomiting (unable to keep anything down)
* Convulsions during present illness
* Lethargic or unconscious state
* Unable to sit or stand up
* Respiratory distress
* Jaundice (observation) or dark urine (by history)
* Severe anemia (Hemoglobin < 5 g/dl)
* Hypotension (systolic BP < 80 mm Hg in adults and < 50 mm Hg in children under the age of 5
* Presence of another significant illness or chronic disease
* Known pregnancy (by history)
* History of hypersensitivity to medication used in the test

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-01; Primary Completion 1999-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of pyrimethamine/sulfdoxine (Fansidar) for the treatment of uncomplicated falciparum malaria in the Peruvian Amazon. | 28 days after dose

CONTACTS AND LOCATIONS:
Overall Officials: Alan Magill, MD, Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Naval Medical Research Center Detachment, Lima, Peru

REFERENCES:
- [Result] Magill AJ, Zegarra J, Garcia C, Marquino W, Ruebush TK 2nd. Efficacy of sulfadoxine-pyrimethamine and mefloquine for the treatment of uncomplicated Plasmodium falciparum malaria in the Amazon basin of Peru. Rev Soc Bras Med Trop. 2004 May-Jun;37(3):279-81. doi: 10.1590/s0037-86822004000300015. PMID 15330070
- [Result] Huaman MC, Roncal N, Nakazawa S, Long TT, Gerena L, Garcia C, Solari L, Magill AJ, Kanbara H. Polymorphism of the Plasmodium falciparum multidrug resistance and chloroquine resistance transporter genes and in vitro susceptibility to aminoquinolines in isolates from the Peruvian Amazon. Am J Trop Med Hyg. 2004 May;70(5):461-6. PMID 15155976
- [Derived] Bacon DJ, Tang D, Salas C, Roncal N, Lucas C, Gerena L, Tapia L, Llanos-Cuentas AA, Garcia C, Solari L, Kyle D, Magill AJ. Effects of point mutations in Plasmodium falciparum dihydrofolate reductase and dihydropterate synthase genes on clinical outcomes and in vitro susceptibility to sulfadoxine and pyrimethamine. PLoS One. 2009 Aug 26;4(8):e6762. doi: 10.1371/journal.pone.0006762. PMID 19707564